CLINICAL TRIAL: NCT05821036
Title: Examining the Effects of Activity Management in Women With Fibromyalgia Syndrome :Randomized Controlled Study
Brief Title: Examining the Effects of Activity Management in Women With Fibromyalgia Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Sena Albay, Research Assistant, Ankara Medipol University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SAlbay
Record Dates: First submitted 2023-03-20; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; activity management; pain management; occupational balance; occupational performance; occupational therapy
MeSH Terms: conditions — Fibromyalgia; Agnosia

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Inclusion criteria:
  * Having been diagnosed with FMS by a specialist physician,
  * Being a woman between the ages of 18-64,
  * To be literate,
  * Having and actively using a smartphone or a computer
  Exclusion criteria:
  * Any disease accompanying FMS, the presence of psychiatric illness and endocrine disorders,
  * Have previous activity management training,
  * Currently and up to 4 weeks on psychotropic medication,
  * Breastfeeding and pregnancy
  Interventions: Behavioral: Activitiy Management
- Control group (No Intervention): Inclusion criteria:
  * Having been diagnosed with FMS by a specialist physician,
  * Being a woman between the ages of 18-64,
  * To be literate,
  * Having and actively using a smartphone or a computer
  Exclusion criteria:
  * Any disease accompanying FMS, the presence of psychiatric illness and endocrine disorders,
  * Have previous activity management training,
  * Currently and up to 4 weeks on psychotropic medication,
  * Breastfeeding and pregnancy

INTERVENTIONS:
Behavioral: Activitiy Management — Activity Management training will be applied for 5 weeks, 2 sessions per week, and the 1st and 10th sessions will be pre and post-training evaluation, a total of 10 individual, internet-based sessions.
  Week 1:Awareness training and ergonomics training including spine anatomy, correct posture use, ergonomic strategies were planned to increase awareness about FMS. Week 2:Focusing on the challenging activities stated by the individuals, it is aimed to change the behavior by arranging the activity resting cycle in daily life. In addition, the management, adaptation and modification of the activities will be provided within the scope of time management training. Week 3: Joint and energy conservation principles training will be given and it is aimed to create body mechanics and proper posture suitable for activities.Week 4: Relaxation training will be provided as a method of coping with pain.Week 5: Re-evaluation/review of the targets set to reduce pain during activities will be provided.
  Arms: Intervention group

SUMMARY:
Purpose: To determine the effects of activity management training on pain, occupational performance, quality of life, depression, anxiety and occupational balance in women with fibromyalgia syndrome (FMS).

In addition to, reducing pain, which is the main symptom of FMS, by regulating the activity-rest cycle, it is aimed to increase people's participation in daily life and improve their quality of life.

Method: A randomized controlled trial. A total of 10 sessions of individual-internet-based activity management training are applied to women with FMS in the intervention group, 2 sessions a week for 5 weeks, 1st and 10th sessions are pre- and post-training evaluation. Assessments before and after training The Revised Fibromyalgia Impact Questionnaire (FIQR), Canadian Occupational Performance Measure(COPM), Pain-activity patterns scale (Pomp/APPS) ,Nottingham Health Profile,The hospital anxiety and depression scale,The Occupational Balance Questionnaire (OBQ) is applied.Although no intervention is applied to the control group, only preliminary and final evaluations are completed.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with FMS by a specialist physician,
* Being a woman between the ages of 18-64,
* To be literate,
* Having and actively using a smartphone or a computer

Exclusion Criteria:

* Any disease accompanying FMS, the presence of psychiatric illness and endocrine disorders,
* Have previous activity management training,
* Currently and up to 4 weeks on psychotropic medication,
* Breastfeeding and pregnancy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2023-12-27 (Estimated)

PRIMARY OUTCOMES:
The Revised Fibromyalgia Impact Questionnaire (FIQ/RFEA) | 15 minute
  It is a questionnaire that evaluates the limitations and functional impairment in patients with fibromyalgia with a total of 21 questions in three sections: function, general and symptoms. All questions are evaluated on a numerical scale between 0-10. The higher the score obtained from the questionnaire, the higher the disability due to fibromyalgia. Turkish validity and reliability was performed by Ediz et al. on female patients with fibromyalgia. (Cronbach's alpha value is 0.89 for FIQR 1st visit (first assessment) and 0.91 for FIQR 2nd visit (second assessment).)
Canadian Occupational Performance Measurement (COPM) | 20 minute
  It focuses on ocuopational performance in all areas of life, including self-care, leisure, and productivity. It is a person-centered scale created for individuals to analyze and prioritize the factors that limit their participation in ADLs. Turkish cultural adaptation, validity and reliability 2017 (Cronbach Alpha internal consistency coefficient 0.9-1.)
Patterns of Activity Measure" (POAM-P) | 15 minute
  It analyzes the altered activity patterns of individuals with chronic pain while creating their activities. The questionnaire consists of 30 questions and all questions are evaluated on a numerical scale between 0-4. Its Turkish adaptation, validity and reliability were performed by Emine Tunç Süygün on patients with chronic low back/neck pain in 2019. (Cronbach's alpha coefficient is 0.941 for avoidance, 0.917 for overdoing, and 0.940 for regulation.)
Nottingham Health Profile (NSP) | 15 minute
  It consists of 38 questions examining the effects of health problems on different areas of quality of life and 6 sections including physical activity, pain, sleep, social isolation, emotional reactions and energy level. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), emotional reactions (9 items). Each sub-parameter is scored between 0-100. 0 indicates best health, 100 indicates worst health. Turkish validity and reliability of the questionnaire Küçükdeveci, McKenna, Kutlay et al. (2002) by
Hospital anxiety depression scale (HADS) | 15 minute
  Hospital anxiety depression scale (HADS) was developed by Zigmoid and Snaith to examine anxiety and depression in individuals with physical illness. 7 questions of the 14-item scale question anxiety and 7 questions about depression symptoms. assessed on a four-point Likert scale.
  The answers given to the questions are scored between 0-3. The sum of the scores of the odd questions gives the anxiety subscale (HAD-A) score, and the sum of the scores of the even questions gives the depression subscale (HAD-D) score. The lowest score that patients can get from both subscales is 0, and the highest score is 21. The Turkish validity and reliability study of the scale was performed by Aydemir in 1997. (Cronbach's alpha coefficient 0.8525 for anxiety, 0.7784 for depression)
Ocupational Balance Questionnaire (OB-Quest) | 15 minute
  Occupational balance, which is considered to be an important component of health and well-being, is a very important concept in occupational therapy.The concept of 'ocupational balance' is the right amount of the perception that it has the oculation and that it has the right variety between ocuations.Opations and roles in the life cycle, personal factors and ıt has a dynamic structure that changes with external factors. There is a constant transition between ocupational imbalance and balance.The Ocupational Balance Questionnaire (OB-Task) is designed as a standard tool to assess a person's ocupational balance. The questionnaire consists of 10 closed-ended questions. The Turkish validity and reliability were evaluated by Bahadır et al. in 2021. The alpha score of the Turkish OB-Quest Cronbach is 0.645 and it has questionable internal consistency.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No